CLINICAL TRIAL: NCT03018561
Title: Cerebral Oxygenation, Cardiac Output, COGnitive Function, and EXercise in Patients With Metabolic Syndrome, Coronary Heart Disease and Chronic Heart Failure
Brief Title: Brain, Cardiac Hemodynamics and Cognition During Exercise in Subjects With Various Cardiovascular Profiles
Acronym: COGNEX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montreal Heart Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: COGNEX-1
Record Dates: First submitted 2016-12-06; First posted 2017-01-12 (Estimated); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Metabolic Syndrome; Coronary Artery Disease; Heart Failure
MeSH Terms: conditions — Metabolic Syndrome; Coronary Artery Disease; Heart Failure | interventions — Exercise; Neuropsychological Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- aged-gender matched healthy controls (Active Comparator): Healthy subjects: with no MetS and no-documented coronary heart disease (CHD), both males and females, aged>18 years will be included in the study, should they provide written informed consent and have a sufficient initial physical and intellectual capacities allowing an independent daily living.
  Interventions: Other: Exercise and Cognitive testing
- patients with metabolic syndrome (Experimental): Patients with MetS and no-documented CHD, both males and females, aged > 18 years will be included in the study, should they provide written informed consent and have a sufficient initial physical and intellectual capacities allowing an independent daily living. Metabolic syndrome (MetS) will be defined according to recent updated criteria (Alberti et al. 2005):presence of at least three of five criteria, namely abdominal obesity (waist circumference cut-off depending on the recently published ethnic-based variations, triglycerides > 1.70 mmol/l, decreased HDL-cholesterol (< 1.0 mmol/l in men and < 1.3 mmol/l in women), systolic blood pressure > 130 mmHg or diastolic blood pressure > 85 mmHg, and FPG > 5.6 mmol/l.
  Interventions: Other: Exercise and Cognitive testing
- patients with coronary heart disease (Experimental): CHD patients, both males and females, aged > 18 years will be included in the study, should they provide written informed consent and have a sufficient initial physical and intellectual capacities allowing an independent daily living. Moreover, they must have documented CHD (prior myocardial infarction, prior coronary angiography or angioplasty, or documented myocardial ischemia on myocardial scintigraphy).
  Interventions: Other: Exercise and Cognitive testing
- patients with chronic heart failure (Experimental): Patients with documented stable chronic heart failure will be recruited if they show the following inclusion criteria:
  * ≥18 years
  * Left ventricular ejection fraction (LVEF) <40% (measured within 6 months of their enrolment by a multigated acquisition Scan, echo or radiological ventriculography)
  * NYHA functional class I-III
  * Optimal therapy at stable doses including a beta-blocker and an ACE inhibitor or ARA for at least 6 weeks prior to investigation (unless documented rationale for variation).
  * Able to perform an symptom limited exercise test.
  * Capacity and willingness to sign the informed consent form.
  Interventions: Other: Exercise and Cognitive testing

INTERVENTIONS:
Other: Exercise and Cognitive testing — Maximal cardiopulmonary test Rest cognitive testing

SUMMARY:
People with cardiovascular risk (CV) factors (obesity, diabetes, etc...) or established heart disease (such as coronary heart disease or chronic heart failure) often have cognitive dysfunction as compared to people without CV risk factors or heart disease. Among the mechanisms, a reduced cardiac output and cerebral blood flow in those people have been suggested. The aim of this study was to compare resting cognitive function, maximal cardiopulmonary function, cardiac output and cerebral hemodynamics during exercise in patients with metabolic syndrome, coronary heart disease, or heart failure vs. healthy subjects.

DETAILED DESCRIPTION:
All subjects will underwent a baseline evaluation including a medical history, physical examination with measurement of height and weight, body composition and fasting blood sample. All subjects will performed a cognitive testing at rest and a maximal cardiopulmonary exercise test (CEPT) with gas exchange analysis. During CEPT, cerebral oxygenation (measured by near-infra red spectroscopy) and cardiac hemodynamics responses (impedance cardiography) will be measured continuously.

ELIGIBILITY:
Inclusion Criteria

* Healthy subjects: with no MetS and no-documented CHD, both males and females, aged>18 years will be included in the study, should they provide written informed consent and have a sufficient initial physical and intellectual capacities allowing an independent daily living.
* Patients with MetS and no-documented CHD, both males and females, aged > 18 years will be included in the study, should they provide written informed consent and have a sufficient initial physical and intellectual capacities allowing an independent daily living. MetS will be defined according to recent updated criteria (Alberti et al. 2005):presence of at least three of five criteria, namely abdominal obesity (waist circumference cut-off depending on the recently published ethnic-based variations, triglycerides > 1.70 mmol/l, decreased HDL-cholesterol (< 1.0 mmol/l in men and < 1.3 mmol/l in women), systolic blood pressure > 130 mmHg or diastolic blood pressure > 85 mmHg, and FPG > 5.6 mmol/l.
* CHD patients, both males and females, aged > 18 years will be included in the study, should they provide written informed consent and have a sufficient initial physical and intellectual capacities allowing an independent daily living. Moreover, they must have documented CHD (prior myocardial infarction, prior coronary angiography or angioplasty, or documented myocardial ischemia on myocardial scintigraphy).
* Patients with documented stable chronic heart failure will be recruited if they show the following inclusion criteria:

  * ≥18 years
  * Left ventricular ejection fraction (LVEF) <40% (measured within 6 months of their enrolment by MUGA Scan, echo or radiological ventriculography)
  * NYHA functional class I-III
  * Optimal therapy at stable doses including a beta-blocker and an ACE inhibitor or ARA for at least 6 weeks prior to investigation (unless documented rationale for variation).
  * Able to perform an symptom limited exercise test.
  * Capacity and willingness to sign the informed consent form.

Exclusion criteria

For healthy subjects:

* lack of expressed written consent
* metabolic syndrome
* coronary heart disease
* chronic systolic heart failure
* resting left ventricular ejection fraction < 40 %
* symptomatic aortic stenosis
* chronic atrial fibrillation
* malignant exertional arrhythmias
* non-cardiopulmonary limitation to exercise (e.g: arthritis or claudication)
* severe exercise intolerance.

For patients with MetS:

* lack of expressed written consent
* coronary heart disease
* chronic systolic heart failure
* resting left ventricular ejection fraction < 40 %
* symptomatic aortic stenosis
* chronic atrial fibrillation
* malignant exertional arrhythmias
* non-cardiopulmonary limitation to exercise (e.g: arthritis or claudication)
* severe exercise intolerance.

For patients with CHD

* lack of expressed written consent
* recent acute coronary event (< 3 months)
* chronic systolic heart failure
* resting left ventricular ejection fraction < 40 %
* symptomatic aortic stenosis
* severe non-revascularizable coronary disease including left main coronary stenosis
* patient awaiting coronary artery bypass surgery
* chronic atrial fibrillation
* presence of permanent ventricular pacemaker
* malignant exertional arrhythmias
* non-cardiopulmonary limitation to exercise (e.g: arthritis or claudication)
* severe exercise intolerance.

For CHF patients:

* Any relative or absolute contraindications to exercise training among patients with stable chronic heart failure according to current recommendations (Working Group on Cardiac Rehabilitation 2001)
* Fixed-rate pacemaker or ICD devices with heart rate limits set lower than the exercise training target heart rate.
* Major cardiovascular event of procedure within the 3 months preceding enrolment in the study.
* Atrial fibrillation
* Heart failure secondary to significant uncorrected primary valvular disease (except for mitral regurgitation secondary to LV dysfunction)
* Heart failure secondary to congenital heart disease or obstructive cardiomyopathy.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2011-01; Primary Completion 2018-01-15 (Actual); Study Completion 2018-01-15 (Actual)

PRIMARY OUTCOMES:
Cerebral hemodynamics measured with near-infra red spectroscopy (NIRS) | Measured within 2 weeks
  Total haemoglobin (ΔtHb): index of brain perfusion (in µM) measured during maximal exercise test.

SECONDARY OUTCOMES:
Resting cognitive function (assessed by the battery test) | Measured within 2 weeks
  Resting cognitive function : will be evaluated by a validated paper-and-pencil full neuropsychological battery test that include: - D-KEFS Color-Word Interference Stroop test : time (sec.)

CONTACTS AND LOCATIONS:
Overall Officials: Anil Nigam, M.D, Principal Investigator — Montreal Heart Institute

IPD SHARING:
Plan to Share IPD: No
no IPD plan